CLINICAL TRIAL: NCT03216850
Title: Alterations of Glycocalyx in Critical Illness and During Major Surgery and Approaches for Glycocalyx Protection. Effect of Parenteral Nutrition and Plasma Lipidome on GCX
Brief Title: Evaluation of Lipid Emulsion on GCX in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Vladimir Cerny, Clinical Professor, University Hospital Hradec Kralove
Other Study IDs: AZVCR 9307_5/a
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in ICU requiring parenteral nutrition
  Interventions: Device: Sublingual microcirculation assessment

INTERVENTIONS:
Device: Sublingual microcirculation assessment — Non-invasive investigation of the endothelial glycocalyx in the sublingual microcirculation.

SUMMARY:
Characterisation of the lipidome and parenteral nutrition modulate the endothelial glycocalyx.

The aim of the study A is to detect any influence of the lipid emulsion on the endothelial glycocalyx in patients in critical care. The targeted cohort is patients on ICU with an indication for parenteral nutrition including lipid emulsion. 15 patients are planned to be enrolled.

Monitored variables: demographic data, type of the population, type of the lipid emulsion, selected variables of the lipid metabolism, sublingual microcirculation (SDF imaging),

ELIGIBILITY:
Inclusion Criteria:

* patients in ICU
* indication for lipid administration as a part of TPN

Exclusion Criteria:

* shock or clinical/laboratory signs of tissue hypoperfusion
* previous lipid infusions (within 3 months before entering study)
* hyperlipidaemia
* hyperglycaemia (over 10 mmol/l)
* current or previous (within 72 hours before entering the study) use of propofol
* pancreatitis
* severe liver failure
* current use of statins

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion criteria admitted to the ICU.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Cerny, MD, Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Třebeš, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients in ICU Requiring Parenteral Nutrition
Started | 15
Completed | 9 (6 patients did not complete the study because of the pre-analytical error.)
Not Completed | 6
Not completed — Pre-analytical error | 6

BASELINE CHARACTERISTICS:
Arm/Group | Patients in ICU Requiring Parenteral Nutrition
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 15
PBR value [Median (Inter-Quartile Range); unit: micrometer] — Perfused Boundary Region (PBR) is an indirect assessment of the endothelial glycocalyx thickness in sublingual microcirculation.
  micrometer | 2.10 [1.97 to 2.33]

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Glycocalyx Thickness
Description: Endothelial glycocalyx thickness was measured indirectly by PBR, which is a lateral movement of the red blood cells from the median column in the microcirculation in micrometers. The higher the PBR is the more damaged the endothelial glycocalyx is.
Time Frame: One week within the ICU care
Measure: Median (Inter-Quartile Range); unit: micrometer
Arm/Group | Patients in ICU Requiring Parenteral Nutrition
Number analyzed (Participants) | 9
micrometer | 2.28 [2.11 to 2.45]

ADVERSE EVENTS:
Description: Measurement of the endothelial glycocalyx thickness is harmless and partially non-invasive. The study was observational and did not aim at collecting the data about adverse events.
Arm/Group | Patients in ICU Requiring Parenteral Nutrition
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03216850/Prot_SAP_000.pdf